CLINICAL TRIAL: NCT03433261
Title: Ketogenic Diet for Reduction of Oxygen Toxicity in Working Divers
Brief Title: Ketogenic Diet for Reduction of CNS Oxygen Toxicity in Working Divers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00070499
Record Dates: First submitted 2018-01-29; First posted 2018-02-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: CNS Oxygen Toxicity, Ketogenic Diet
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Each subject will randomize to one of two arms and will crossover to the other arm at least one week later.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neither the investigator nor the outcomes assessor will no the ketone level of the participant during either arm of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Diet (No Intervention): The participant will eat their usual diet for at least 72 hrs prior to the experiment, document their diet during that time and be tested for ketone level immediately prior to the experiment.
- Ketogenic Diet (Experimental): The participant will follow a ketogenic diet for 72 hrs prior to the experiment and consume a ketone supplement 60 minutes prior to the experiment. They will document their diet and be tested for ketone level immediately prior to the experiment.
  Interventions: Dietary Supplement: Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — Eat a ketogenic diet (low carbohydrate, high fat diet) for 72 hrs prior to the experiment and consume a dietary ketone supplement 60 minutes before the experiment.
  Arms: Ketogenic Diet

SUMMARY:
The purpose of this research study is to understand the effect of nutritional ketosis on CNS oxygen toxicity in undersea divers. The investigators hope this will provide a starting point to develop methods for improving the safety of Navy divers, warfighters and submariners.

DETAILED DESCRIPTION:
Participants in the study will undergo a physical exam and testing as well as training on cognitive testing software as part of the screening process. Eligible subjects will be assigned a normal diet or a ketogenic diet (a diet high in fat/protein and low in carbohydrates) for three days before testing. Subjects will be immersed in water to the shoulders, inside a hyperbaric (high pressure) chamber while breathing 100% oxygen at increased atmospheric pressure, and doing cycling exercise. Testing on the cognitive software, as well as blood sampling and physical monitoring will be done while in the chamber. All tests and procedures will be completed again at least one week later with the diet not assigned for the first session.

ELIGIBILITY:
Inclusion Criteria:

* Males & females between 18 and 50 years old
* Able to pedal a bicycle ergometer continuously for 15 minutes
* Non-smoker
* No history of cardiovascular disease, including coronary artery disease, valvular disease, cardiomyopathy or hypertension.
* No history of lung disease

Exclusion Criteria:

* Prolonged QTc on initial ECG
* Currently pregnant or attempting to become pregnant.
* Have a history of:

  1. Smoking
  2. Coronary artery disease
  3. Hypertension
  4. Seizures
  5. Exercise intolerance
  6. Psychiatric disorder
  7. Previous pneumothorax or pneumomediastinum
  8. Hypo or hyperglycemia
  9. Diabetes
* Regularly take any medications which may alter heart rate, blood pressure, neurotransmitter function, mood or affect.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Time to First Manifestations of CNS Oxygen Toxicity | 2 hrs
  Time to the first manifestation of CNS Oxygen Toxicity: visual or hearing changes, nausea, twitching, irritability, dizziness, convulsions or change consistent with possible CNS Oxygen Toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No